CLINICAL TRIAL: NCT03207360
Title: Pain Coping Skills Training and Meaning-Centered Intervention for Cancer Pain
Brief Title: Pain Coping Skills and Meaning-Centered Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083582; 130526-PF-17-054-01-PCSM (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancer; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Coping Skills (Experimental)
  Interventions: Behavioral: Pain Coping Skills

INTERVENTIONS:
Behavioral: Pain Coping Skills — Participants will be trained in pain coping skills and meaning-centered psychotherapy. The intervention will consist of 4 weekly videoconference-delivered sessions that will last between 45 and 60 minutes.
  Other Names: Meaning-Centered Psychotherapy

SUMMARY:
The proposed study seeks to develop and test a novel psychosocial pain management intervention for patients with advanced cancer. It is hypothesized that the intervention will demonstrate feasibility, acceptability, and preliminary efficacy. The first aim is to develop a combined pain coping skills training and meaning-centered psychotherapy intervention. The second aim is to test the intervention's feasibility and acceptability as well as preliminary efficacy for improving primary outcomes (i.e., pain, pain interference, and meaning in life) and secondary outcomes. Two efficacious, theory-driven interventions will be integrated to address pain management by teaching pain coping skills with a novel emphasis on enhancing a sense of meaning in life. Participants will be patients with advanced cancer and moderate-to-severe pain. The study will be conducted in two phases. Phase I of the study will be intervention development. The intervention content will be guided by theory and mentoring from a team of leading experts in pain management and meaning-centered psychotherapy. Initial intervention content will be further informed by interviews with patients with advanced cancer. Content will then be refined through an iterative patient testing process. Phase II of the study will be a single-arm pilot trial testing the intervention. The intervention will be delivered in-person and consist of four, 45-to-60 minute therapy sessions delivered using videoconferencing technology. Study measures will be collected at baseline (0 weeks), immediately post-intervention (5 weeks), and 4-weeks post-intervention (9 weeks).

DETAILED DESCRIPTION:
Effective pain management is a major healthcare concern for patients with advanced cancer. Compared to patients with early-stage disease, those with advanced cancer report higher levels of pain and greater functional impairment related to pain. There is a critical need for psychosocial pain management interventions that are specifically designed to address the suffering of patients with advanced cancer. The proposed study seeks to develop and assess the feasibility, acceptability, and preliminary efficacy of a novel integration of pain coping skills training and meaning-centered psychotherapy for patients with advanced cancer and moderate-to-severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV solid tumor cancer diagnosis; or stage III pancreatic or lung cancer diagnosis
* At least moderate pain (pain score >/= 4) at recruitment
* Clinically elevated distress (NCCN Distress Thermometer >/= 3) at recruitment
* Eastern Cooperative Oncology Group (ECOG) </= 2 at recruitment
* Ability to speak and read English

Exclusion Criteria:

* Brain tumor diagnosis
* Significant cognitive impairment
* Serious mental illness that would interfere with engagement in the intervention (e.g., schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by study accrual | 5 weeks (immediately post-intervention)
  Treatment feasibility will be shown by meeting targeted study accrual (N = 30 for single-arm trial) in the 24-month study period.
Feasibility as measured by study attrition | 5 weeks (immediately post-intervention)
  Treatment feasibility will be shown by no more than 30% study attrition. Attrition will be defined as not completing the post-intervention assessment.
Acceptability as measured by the Client Satisfaction Questionnaire eight-item version (CSQ) | 5 weeks (immediately post-intervention)
  Acceptability will be indicated by at least 80% of the participants reporting satisfaction with the protocol (mean score of 7) on the CSQ.
Acceptability as measured by engagement | 3 weeks, 4 weeks, and 5 weeks (sessions 2, 3, and 4)
  Acceptability will be indicated by reported practice of the skills and ideas from the intervention in at least 75% of the sessions.
Change in pain and pain interference | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Pain and pain interference will be measured using the 11-item Brief Pain Inventory-Short Form (BPI-SF).
Change in meaning in life | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Meaning in life (i.e., purpose, coherence, and significance) and overall spiritual well-being will be measured using the 12-item Functional Assessment of Cancer Therapy - Spiritual Well-Being scale (FACIT-Sp).

SECONDARY OUTCOMES:
Change in self-efficacy for pain management | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Self-efficacy for pain management will be measured using the five-item self-efficacy for pain management subscale of the Chronic Pain Self-Efficacy Scale.
Change in anxiety | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Anxiety will be measured using the seven-item version of the Generalized Anxiety Disorders scale (GAD-7).
Change in depressive symptoms | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Depressive symptoms will be measured using the eight-item version of the Patient Health Questionnaire (PHQ-8).
Change in hopelessness | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Hopelessness will be measured using the eight-item Hopelessness Assessment in Illness Questionnaire.
Change in fatigue | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Fatigue will be assessed using the four-item Fatigue Symptom Inventory (FSI).
Change in health-related quality of life | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Health-related quality of life will be assessed using the 16-item version of the McGill Quality of Life Questionnaire.
Change in performance status | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Performance status will be assessed using the one-item self-report version of the Karnofsky Performance Rating Scale.
Change in meaningfulness in life despite pain | 0 weeks, 5 weeks, and 9 weeks (baseline, immediately post-intervention, 4-weeks post-intervention)
  Meaningfulness in life despite pain will be measured using the five-item Pain Solutions Questionnaire - Meaningfulness in Life Despite Pain subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G Winger, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winger JG, Ramos K, Kelleher SA, Somers TJ, Steinhauser KE, Porter LS, Kamal AH, Breitbart WS, Keefe FJ. Meaning-Centered Pain Coping Skills Training: A Pilot Feasibility Trial of a Psychosocial Pain Management Intervention for Patients with Advanced Cancer. J Palliat Med. 2022 Jan;25(1):60-69. doi: 10.1089/jpm.2021.0081. Epub 2021 Aug 12. PMID 34388037